CLINICAL TRIAL: NCT06816316
Title: Role of Alcohol in Prevention of Recurrence of the Accidentally Opened Angular Dermoid Cyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohamed Yasser Sayed Saif, Dean of National Institute of Longevity Elder Sciences - Professour of Ophthalmology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMBSUREC/01102024/Saeed
Record Dates: First submitted 2024-04-28; First posted 2025-02-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Dermoid Cyst; Choristomas
Keywords: dermoid cyst; ethyl alcohol; choristomas; lipogranulomatous inflammatory
MeSH Terms: conditions — Dermoid Cyst; Choristoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) (Placebo Comparator): only saline was used to wash the surgical field
  Interventions: Procedure: external angular dermoid cysts surgical removal
- group (B) (Active Comparator): ethyl alcohol 70% was used to wash the surgical field
  Interventions: Procedure: external angular dermoid cysts surgical removal

INTERVENTIONS:
Procedure: external angular dermoid cysts surgical removal — Skin incision was done below the eyebrow, subcutaneous and orbicularis dissection was done to remove the cysts. Upon accidental opening of the cyst then removal of the cyst walls and its contents from the surgical field as much as possible was done.
  At this step, in group (A) only saline was used to wash the surgical field from any remnants. In group (B) the surgical field was cleaned with a gauze soaked with ethyl alcohol 70%. Then closure of the wound in both groups.

SUMMARY:
Purpose to evaluate the effect of alcohol used in accidentally opened dermoid cyst in prevention of inflammation and recurrence Patient and method: Itt is a comparative interventional study ,performed on 60 patients with external angular dermoid cysts that were accidentally opened during surgical removal , they were divided into two groups ,Group (A) includes 30 patients where only saline was used to wash the surgical field while group(B) includes 30 patients where ethyl alcohol 70% was used.

DETAILED DESCRIPTION:
1. Study Design and Rationale:

   This is a comparative interventional study designed to evaluate the efficacy of 70% ethyl alcohol in preventing inflammation and recurrence in cases of accidentally opened external angular dermoid cysts during surgical removal. The rationale for using 70% ethyl alcohol is based on its antimicrobial and antiseptic properties, which may reduce the risk of postoperative infection and cyst recurrence compared to saline irrigation alone.
2. Patient Recruitment and Group Allocation:

   Recruitment Sites: Patients were recruited from outpatient clinics at Beni-Suef University Hospitals, Fayoum University Hospitals, and MUST University Hospital.

   Recruitment Period: May 2022 to May 2024.

   Group Allocation:

   Group A (Control Group): 30 patients treated with saline irrigation.

   Group B (Intervention Group): 30 patients treated with 70% ethyl alcohol.
3. Surgical Procedure:

   Preoperative Preparation:

   Patients were positioned supine, and the surgical site was sterilized using standard antiseptic protocols.

   Local or general anesthesia was administered based on patient and surgeon preference.

   Incision and Dissection:

   A skin incision was made below the eyebrow, followed by subcutaneous and orbicularis dissection to expose the dermoid cyst.

   Care was taken to avoid accidental rupture, but if the cyst was opened, the following steps were implemented.

   Cyst Management:

   The cyst walls and contents were meticulously removed from the surgical field to minimize residual material.

   Group A (Saline Group): The surgical field was irrigated with sterile saline solution to remove any remnants.

   Group B (Alcohol Group): The surgical field was cleaned using a gauze soaked with 70% ethyl alcohol to ensure thorough disinfection.

   Wound Closure:

   The wound was closed in layers using absorbable sutures for subcutaneous tissues and non-absorbable sutures or skin adhesive for the skin.

   A sterile dressing was applied.
4. Postoperative Care:

   Medications:

   Both groups received the same regimen of systemic antibiotics (e.g., amoxicillin-clavulanate) and anti-inflammatory drugs (e.g., ibuprofen) for 5-7 days to prevent infection and inflammation.

   Follow-Up:

   Patients were monitored at 1 week, 1 month, 3 months, and 6 months postoperatively.

   At each visit, the surgical site was assessed for signs of inflammation, infection, or recurrence.

   Any adverse events or complications were recorded.
5. Data Collection and Analysis:

   Data Collected:

   Demographic data (age, sex).

   Intraoperative details (cyst size, extent of spillage).

   Postoperative outcomes (infection, inflammation, recurrence).

   Statistical Methods:

   Data were analyzed using SPSS version 24.

   Quantitative variables (e.g., cyst size) were summarized as mean ± standard deviation.

   Categorical variables (e.g., recurrence rates) were summarized as frequencies and percentages.

   Comparisons between groups were performed using:

   ANOVA with post hoc tests for continuous variables.

   Chi-square test or Fisher's exact test for categorical variables.

   Pearson correlation coefficient was used to assess relationships between quantitative variables.

   A p-value < 0.05 was considered statistically significant.
6. Technical Considerations:

   Ethyl Alcohol Concentration: 70% ethyl alcohol was chosen for its optimal balance between antimicrobial efficacy and tissue safety.

   Saline Irrigation: Sterile saline was used as a control to mimic standard surgical practice.

   Standardization: All procedures were performed by experienced surgeons to ensure consistency in technique and cyst management.
7. Ethical and Regulatory Compliance:

   Informed Consent: Written informed consent was obtained from all participants prior to surgery.

   Ethical Approval: The study protocol was approved by the Ethics Committee of Beni-Suef University and adhered to the principles of the Helsinki Declaration.

   Patient Safety: Adverse events were monitored and managed promptly to ensure patient safety.
8. Limitations:

   The study is limited by its sample size (n=60), which may affect the generalizability of the results.

   The follow-up period of 6 months may not be sufficient to capture long-term recurrence rates.

   Potential variability in surgical technique among different surgeons.
9. Expected Outcomes:

The study aims to demonstrate that 70% ethyl alcohol is more effective than saline in reducing postoperative inflammation and recurrence in accidentally opened dermoid cysts.

If proven effective, this intervention could be incorporated into standard surgical protocols for dermoid cyst management.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of external angular dermoid cyst.

Accidental opening of the dermoid cyst during surgical removal.

Age: Patients of any age eligible for surgical intervention.

Willingness to provide written informed consent for participation in the study.

Exclusion Criteria:

Recurrent dermoid cysts (previously treated or excised).

Complicated dermoid cysts (e.g., preoperatively ruptured or infected).

Patients with contraindications to the use of ethyl alcohol (e.g., known hypersensitivity or allergy).

Patients with systemic conditions that may impair wound healing (e.g., uncontrolled diabetes, immunocompromised states).

Patients who are pregnant or breastfeeding.

Patients unable or unwilling to comply with follow-up visits.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
post-operative inflammation | 6 month
  The primary outcome of post-operative inflammation measures the incidence of clinically significant inflammatory responses at the surgical site following excision of an accidentally opened external angular dermoid cyst. Inflammation is defined as the presence of two or more of the following clinical signs:
  Erythema (redness) extending ≥1 cm from the wound edges.
  Edema (swelling) at or around the surgical site.
  Local warmth compared to adjacent skin.
  Pain or tenderness reported by the patient or elicited during palpation.
  Purulent discharge from the incision site.

SECONDARY OUTCOMES:
recurrence | 6 month
  The recurrence outcome measures the number of participants who experience a reappearance of the external angular dermoid cyst at the surgical site within the 6-month follow-up period after surgical removal. Recurrence is defined as the presence of a palpable mass or radiologically confirmed lesion (via ultrasound or MRI) that exhibits characteristics consistent with a dermoid cyst. This outcome is a critical measure of the long-term efficacy of the surgical intervention and the intraoperative cleaning method (saline vs. 70% ethyl alcohol) in preventing residual cyst material from causing regrowth.

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Fayoum University Hospital, Al Fayyum, Faiyum Governorate
  - Beni Suef University, Banī Suwayf
  - Misr University For Science and Technology, Giza

IPD SHARING:
Plan to Share IPD: No